CLINICAL TRIAL: NCT06535555
Title: Safety and Feasibility of ActivSight(tm) in the Identification of The Ureter Via Riboflavin Fluorescence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was never initiated.
Sponsor: Activ Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 600-00012
Record Dates: First submitted 2023-02-10; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Surgical Procedure, Unspecified
Keywords: ureter, advanced imaging, surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Investigational Arm (Experimental): Patients in the investigational arm will ingest 400mg PO riboflavin pre-operatively. At the start of their procedure, after the surgeon gain laparoscopic access using their standard procedures and equipment, the updated version of the ActivSight device will be placed through a standard laparoscopic trocar and attempts will be made to visualize the ureter under direct imaging using light in the visible spectrum.
  When the surgeon is complete with the attempted visualization, they will remove the ActivSight device and proceed with their normal operative course and equipment.
  No surgical decisions will be made based upon this information, and the device will only be used during the aforementioned time.
  Interventions: Device: Investigational Safety and Feasibility

INTERVENTIONS:
Device: Investigational Safety and Feasibility — Technical feasibility will be assessed based on a five-point rating scale assessing the ease-of-use, ureteral visibility, and time required to identify the ureter using ActivSight™. All images and video of the ureter will be recorded, but surgeon feedback will be used to assess technical success based on a five point scale, rather than these (subsequently de-identified) recordings.
  Safety will be confirmed through clinical assessments and evaluation of adverse events intraoperatively and through a 28-day follow-up period using the criteria listed below. All adverse events will be adjudicated by the site's Principal Investigator (PI) to judge the relatedness of the adverse event to either the administration of riboflavin or the use of the prototype ActivSight™ device (or whether the adverse event was unrelated to either)

SUMMARY:
The main Objective of this study is to determine the safety and feasibility of a prototype ActivSightTM in identifying the ureter in real-time during elective laparoscopic abdominopelvic surgery after pre-surgical administration of riboflavin. This study seeks to identify the ureter only; ActivSight™ will not be used to Safety and Feasibility of ActivSightTM in the Identification of the Ureter via Riboflavin Fluorescence guide treatment or the surgical procedure. As such, this is a non-significant risk study. Riboflavin is a common dietary supplement and will be administered at dosages shown previously to be well-tolerated for migraine prophylaxis [6]. ActivSight™ is an imaging system connected to the standard laparoscopic system already existing in the OR at the site. Changes made to the commercial ActivSight™ hardware for this study introduce no significant risk

DETAILED DESCRIPTION:
In the 2019 publication, "A zwitterionic near-infrared fluorophore for real-time ureter identification during laparoscopic abdominopelvic surgery," by de Valk, et al. [1], the authors present the clinical need for real-time identification of the ureter during laparoscopic abdominal surgery: "Iatrogenic ureteral injury is amongst the most feared complications of lower abdominal surgery, with incidence varying from 0.5 - 1% in cancer surgery, to as high as 10% in gynecologic oncologic surgery [2-5]. Ureters are thin-walled and at risk for injury as they are poorly distinguished from surrounding retroperitoneal tissue and are usually in a collapsed state. Unrecognized ureteral damage during surgery can lead to long-term morbidity, including kidney failure." In their publication, this team proposes the use of a zwitterionic near-infrared fluorophore that could be detected in real-time via near-infrared fluorescence imaging. Activ Surgical has developed and commercialized ActivSight™, a near-infrared fluorescence detector, that combines an innovative form factor and proprietary software to deliver precise, objective, cost efficient real-time visualization of blood flow and tissue perfusion intraoperatively for laparoscope-based surgery. A small adaptor fits between any existing laparoscope and camera system and a separate light source is placed along any current commercial system to deliver objective real-time tissue perfusion and blood flow information intraoperatively. ActivSight™ received 510(k) clearance from the US FDA in 2020. According to its labelling, ActivSight™ is intended to provide real-time endoscopic fluorescence and near infrared imaging. ActivSight™ enables surgeons to visually assess blood flow and related tissue perfusion using fluorescence and near infrared imaging, and at least one of the major bile ducts (cystic duct, common bile duct or common hepatic duct) using fluorescence, all during minimally invasive surgery. In this clinical feasibility study, Activ Surgical proposes a slightly different approach from the above-referenced publication to achieve real-time ureter identification during elective laparoscopic abdominal surgery. Instead of utilizing a zwitterionic fluorophore to fluoresce the ureter, Activ Surgical is investigating a common over-the-counter water-soluble vitamin: riboflavin, also known as vitamin B2.

While typically administered as a dietary supplement, the medical literature contains many large studies of riboflavin use as prophylaxis for migraines [6]. It has also been studied and used to identify ureteral jets during cystoscopy as a method of confirming ureter patency after pelvic prolapse surgery [7-8].

Riboflavin possesses properties of fluorescence, with three strong areas of fluorescence [9] in the visible wavelength spectrum. To detect the fluorescence of riboflavin, changes were made to ActivSight™ hardware for this study; these changes are detailed herein. The main Objective of this study is to determine the safety and feasibility of a prototype ActivSightTM in identifying the ureter in real-time during elective laparoscopic abdominopelvic surgery after pre-surgical administration of riboflavin. This study seeks to identify the ureter only; ActivSight™ will not be used to guide treatment or the surgical procedure. As such, this is a non-significant risk study. Riboflavin is a common dietary supplement and will be administered at dosages shown previously to be well-tolerated for migraine prophylaxis [6]. ActivSight™ is an imaging system connected to the standard laparoscopic system already existing in the OR at the site. Changes made to the commercial ActivSight™ hardware for this study introduce no significant risk. Subjects presenting for elective laparoscopic abdominopelvic surgery (meeting the inclusion/exclusion criteria detailed below) will be consented and asked to permit the surgeons to identify their ureter with the prototype ActivSight™ system during elective laparoscopic surgery after ingesting the proper dosage of riboflavin pre-surgery. Video of the ureter examination will be recorded and analyzed post-surgery; retained video will be devoid of any protected health information.

ELIGIBILITY:
Inclusion Criteria:

* Ages 22 to 65 presenting for elective laparoscopic abdominopelvic surgery
* No contraindication to riboflavin and able to ingest riboflavin in pill form
* Willing and able to consent to the study
* Native language is English or proficient in both written and spoken English

Exclusion Criteria:

* Known or suspected history of any of the following:

  * Kidney or liver disease
  * Vitamin deficiency or transporter deficiency or metabolic disorder
  * Pelvic surgery (including gynecologic, colorectal, urologic, etc.)
  * Pelvic radiation
  * Abdominopelvic trauma
  * Ureteral injury or presence of ureteral stent(s)
  * Bladder injury
  * Kidney stones
  * Inflammatory bowel disease
  * Neurologic disorder, including seizure or stroke history (history of migraine is acceptable)
  * Any form of diabetes
* Active malignancy
* Uncontrolled hypertension
* Multiple chronic recurring urinary tract infections (isolated urinary tract infections are acceptable)
* BMI > 35 kg/m2
* Pregnant or lactating

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Ureteral visibility | Immediately post-operative
  1-5 point scale, surgeon assessment of how visible the ureter was on imaging
Ease of use | Immediately post-operative
  1-5 point scale, surgeon assessment of how easy the technology was to use intraoperatively
Time required to identify ureter | Immediately post-operative
  1-5 point scale, surgeon assessment of how much time it took to identify the ureter

OTHER OUTCOMES:
Adverse events | 28 days post-op
  Adverse events will be summarized descriptively and tabulations on the type, severity, and relationship to the prototype ActivSight™ or administration of riboflavin will be performed and any changes of outcomes from baseline on follow up will be examined using the nonparametric Wilcoxon rank test.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Special Surgery, Roswell, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Valk KS, Handgraaf HJ, Deken MM, Sibinga Mulder BG, Valentijn AR, Terwisscha van Scheltinga AG, Kuil J, van Esdonk MJ, Vuijk J, Bevers RF, Peeters KC, Holman FA, Frangioni JV, Burggraaf J, Vahrmeijer AL. A zwitterionic near-infrared fluorophore for real-time ureter identification during laparoscopic abdominopelvic surgery. Nat Commun. 2019 Jul 16;10(1):3118. doi: 10.1038/s41467-019-11014-1. PMID 31311922
- [Background] Delacroix SE Jr, Winters JC. Urinary tract injures: recognition and management. Clin Colon Rectal Surg. 2010 Jun;23(2):104-12. doi: 10.1055/s-0030-1254297. PMID 21629628
- [Background] Andersen P, Andersen LM, Iversen LH. Iatrogenic ureteral injury in colorectal cancer surgery: a nationwide study comparing laparoscopic and open approaches. Surg Endosc. 2015 Jun;29(6):1406-12. doi: 10.1007/s00464-014-3814-1. Epub 2014 Aug 26. PMID 25154890
- [Background] Engel O, Rink M, Fisch M. Management of iatrogenic ureteral injury and techniques for ureteral reconstruction. Curr Opin Urol. 2015 Jul;25(4):331-5. doi: 10.1097/MOU.0000000000000175. PMID 26049877
- [Background] Thompson DF, Saluja HS. Prophylaxis of migraine headaches with riboflavin: A systematic review. J Clin Pharm Ther. 2017 Aug;42(4):394-403. doi: 10.1111/jcpt.12548. Epub 2017 May 8. PMID 28485121
- [Background] Fernando S, Dowling C, Rosamilia A. The role of preoperative oral vitamin B in the cystoscopic assessment of ureteric patency. Int Urogynecol J. 2011 Aug;22(8):947-51. doi: 10.1007/s00192-011-1396-1. Epub 2011 Apr 7. PMID 21472446
- [Background] Stitely ML, Harlow K, MacKenzie E. Oral Riboflavin to Assess Ureteral Patency During Cystoscopy: A Randomized Clinical Trial. Obstet Gynecol. 2019 Feb;133(2):301-307. doi: 10.1097/AOG.0000000000003063. PMID 30633139